CLINICAL TRIAL: NCT01146912
Title: TextFluenza: Using Technology To Promote Flu Vaccination In Underserved Maternal And Child Population
Brief Title: TextFluenza: Using Technology To Promote Flu Vaccination In Underserved Maternal And Child Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Asst Prof of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAF0137; R40MC17169-01 (Other Grant/Funding Number: R40MC17169-01)
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-09

CONDITIONS: Influenza
Keywords: Influenza, text message, vaccination
MeSH Terms: conditions — Influenza, Human | interventions — Health Services

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message vaccine reminders (Experimental): Receipt of text message vaccine reminders
  Interventions: Other: Text Message; Other: automated call
- automated phone call from clinic (Active Comparator): Receipt of automated phone call from clinic
  Interventions: Other: automated call

INTERVENTIONS:
Other: Text Message — Text message vaccine reminders
  Other Names: Health services
  Arms: Text message vaccine reminders
Other: automated call — Automated call
  Other Names: Health services

SUMMARY:
The Advisory Committee on Immunization Practices (ACIP)recommends that the flu vaccine be administered annually to all children aged 6 months to 18 years as well as women who are pregnant during the influenza season. Nevertheless, targeting and mobilizing these populations has been difficult and influenza immunization rates nationwide remain low. Immunization reminder-recalls have been shown to be effective, but have had limited ability to rapidly identify and reach large target populations in a cost-effective manner. Evidence on how to optimally design these systems is not yet available and thus text message immunization alerts have not been widely implemented. The investigators propose to implement and evaluate tailored, targeted influenza text message reminders in urban pediatric and pregnant populations.

ELIGIBILITY:
Inclusion criteria Parents (2010-2011 and 2011-2012 influenza seasons)

* Children aged 6 months to 18 years at the beginning of current influenza season
* Children with one previous visit at participating pediatric community health center in last year
* Parent with cell phone number in registry

Pregnant women Pilot (2010-2011 influenza seasons)

* Pregnant women who will be in their 2nd or 3rd trimester during the influenza season
* Own a cell phone with text message capability

Randomized controlled Trial (2011-2012 influenza seasons)

* Pregnant and will be in their 2nd or 3rd trimester during the influenza season
* Cell phone number in registry

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30537 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Stockwell MS, Westhoff C, Kharbanda EO, Vargas CY, Camargo S, Vawdrey DK, Castano PM. Influenza vaccine text message reminders for urban, low-income pregnant women: a randomized controlled trial. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):e7-12. doi: 10.2105/AJPH.2013.301620. Epub 2013 Dec 19. PMID 24354839
- [Derived] Stockwell MS, Kharbanda EO, Martinez RA, Vargas CY, Vawdrey DK, Camargo S. Effect of a text messaging intervention on influenza vaccination in an urban, low-income pediatric and adolescent population: a randomized controlled trial. JAMA. 2012 Apr 25;307(16):1702-8. doi: 10.1001/jama.2012.502. PMID 22535855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children and pregnant women receiving care at 4 community-based clinics in the United States during the 2010-2011, 2011-2012 influenza season
Pre-assignment Details: Children previously vaccinated for influenza before the season of interest were excluded from primary analysis
Groups:
- Pediatric Text Message Vaccine Reminders/Automated Phone Call: Receipt of text message vaccine reminders, in addition to standard of care of automated phone call from clinic
- Pediatric: Automated Phone Call From Clinic Only: Receipt of automated phone call from clinic
- Pregnant Women: Text Message: Received text message reminders
- Pregnant Women: Usual Care: Received usual care
- Delayed Pediatrics: Interactive Text Message Vaccine Reminders: Vaccination of children not yet vaccinated by mid-November: interactive message
- Delayed Pediatric: Conventional Text Message: Vaccination of children not yet vaccinated by mid-November: conventional text message
- Delayed Pediatric: Usual Care: Vaccination of children not yet vaccinated by mid-November: usual care
- Parents: Included in enrollment but not in outcomes which are on child level
Period: Overall Study
Arm/Group | Pediatric Text Message Vaccine Reminders/Automated Phone Call | Pediatric: Automated Phone Call From Clinic Only | Pregnant Women: Text Message | Pregnant Women: Usual Care | Delayed Pediatrics: Interactive Text Message Vaccine Reminders | Delayed Pediatric: Conventional Text Message | Delayed Pediatric: Usual Care | Parents
Started | 4607 | 4606 | 593 | 594 | 1821 | 1821 | 1820 | 14675
Completed | 3790 | 3784 | 576 | 577 | 1780 | 1760 | 1764 | 14675 (Parents are considered subjects but outcomes are on child level)
Not Completed | 817 | 822 | 17 | 17 | 41 | 61 | 56 | 0
Not completed — Already received influenza vaccination | 817 | 822 | 13 | 15 | 41 | 61 | 56 | 0
Not completed — < 14 weeks gestational age | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Duplicate patient | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Text Message Vaccine Reminders/Automated Telephone Call: Receipt of text message vaccine reminders, in addition to standard of care of automated phone call from clinic
- Automated Phone Call From Clinic Only: Receipt of automated phone call from clinic
- Total: Total of all reporting groups
Arm/Group | Text Message Vaccine Reminders/Automated Telephone Call | Automated Phone Call From Clinic Only | Pregnant Women: Text Message | Pregnant Women: Usual Care | Delayed Pediatrics: Interactive Text Message | Delayed Pediatrics: Conventional Text Message | Delayed Pediatrics: Usual Care | Total
Number analyzed (Participants) | 4607 | 4606 | 593 | 594 | 1821 | 1821 | 1820 | 15862
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4607 | 4606 | 0 | 0 | 1821 | 1821 | 1820 | 14675
  Between 18 and 65 years | 0 | 0 | 593 | 594 | 0 | 0 | 0 | 1187
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2335 | 2332 | 593 | 594 | 869 | 926 | 862 | 8511
  Male | 2272 | 2274 | 0 | 0 | 952 | 895 | 958 | 7351
Region of Enrollment [Number; unit: participants]
  United States | 4607 | 4606 | 593 | 594 | 1821 | 1821 | 1820 | 15862

OUTCOME MEASURES:

1. Primary Outcome: Influenza Immunization: Pediatric
Description: percentage of pediatric participants with influenza immunization by March 31 of 2011
Time Frame: March 31, 2011
Population: Individuals unvaccinated by time intervention start for their cohort
Measure: Number; unit: % participant vaccinated with influenza
Groups:
- Pediatric: Text Message Vaccine-reminders/Automated Phone Call: Receipt of text message vaccine reminders, in addition to standard of care of automated phone call from clinic
Arm/Group | Pediatric: Text Message Vaccine-reminders/Automated Phone Call | Pediatric: Automated Phone Call From Clinic Only
Number analyzed (Participants) | 3790 | 3784
% participant vaccinated with influenza | 43.6 | 39.9

2. Secondary Outcome: Pediatric: Vaccinated at Influenza Clinic
Description: percentage of pediatric participants vaccinated at an influenza immunization clinic by March 31 of 2011
Time Frame: March 31, 2011
Population: those unvaccinated by the start date for their cohort
Measure: Number; unit: % participant vaccinated at flu clinic
Groups:
- Pediatric: Text Message Vaccine Reminders/Automated Phone Call: Receipt of text message vaccine reminders, in addition to standard of care of automated phone call from clinic
Arm/Group | Pediatric: Text Message Vaccine Reminders/Automated Phone Call | Pediatric: Automated Phone Call From Clinic Only
Number analyzed (Participants) | 3790 | 3784
% participant vaccinated at flu clinic | 6.1 | 2.8

3. Secondary Outcome: Attendance at Appointment
Description: percentage of pregnant participants who attended an appointment a reminder for from Sept-December 2011
Time Frame: September-December 2011
Measure: Number; unit: % participants attending appointment
Arm/Group | Text Message Vaccine Reminders | Automated Phone Call From Clinic
Number analyzed (Participants) | 576 | 577
% participants attending appointment | 85.0 | 87.6

4. Primary Outcome: Influenza Immunization: Pregnant Women
Description: percentage of pregnant participants with influenza immunization by December 31, 2011
Time Frame: by December 31, 2011
Measure: Number; unit: %participants vaccinated with influenza
Arm/Group | Pregnant Women: Text Message | Pregnant Women: Usual Care
Number analyzed (Participants) | 576 | 577
%participants vaccinated with influenza | 49.3 | 46.6

5. Primary Outcome: Influenza Immunization: Delayed Pediatric
Description: percentage of pediatric participants with influenza immunization by March 31 of 2012
Time Frame: March 31, 2012
Measure: Number; unit: %participants vaccinated with influenza
Arm/Group | Delayed Pediatrics: Interactive Text Message Vaccine Reminders | Delayed Pediatric: Conventional Text Message | Delayed Pediatric: Usual Care
Number analyzed (Participants) | 1780 | 1760 | 1764
%participants vaccinated with influenza | 38.5 | 35.3 | 34.8

ADVERSE EVENTS:
Description: Only Serious Adverse Events were collected/assessed
Arm/Group | Pediatric: Text Message Vaccine-reminders/Automated Phone Call | Pediatric: Automated Phone Call From Clinic Only | Pregnant Women: Text Message | Pregnant Women: Usual Care | Delayed Pediatric: Interactive Text Message | Delayed Pediatric: Conventional Text Message | Delayed Pediatric: Usual Care
Serious Adverse Events (participants affected / at risk) | 0/4607 | 0/4606 | 0/593 | 0/594 | 0/1821 | 0/1821 | 0/1820
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No